CLINICAL TRIAL: NCT02517047
Title: Community Empowerment to Pilot a Novel Device for Monitoring Rescue Medication Use in Urban Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Principle Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P00018778
Record Dates: First submitted 2015-07-27; First posted 2015-08-06 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CareTRx Device (Experimental): Subject will receive CareTRx device for rescue inhaler as well as the application downloaded to their Android phone. The device will track when the rescue inhaler is administered. The information will then be loaded to phone app.
  Interventions: Device: CareTRx

INTERVENTIONS:
Device: CareTRx — CareTRx is a novel device that can be applied to most MDI (meter dose inhaler) device and leverages mobile and cloud computing to objectively assess and provide real-visualize feedback to patients and providers around medication adherence and disease control in pediatric asthma.

SUMMARY:
Background: Pediatric asthma is the most common chronic illness among children and is associated with poor quality of life, activity restriction, school absences, and thousands of physician visits annually. The purpose of this study is to measure the effectiveness of using an innovative tracking system (CareTRx) for the self-management of asthma, including daily and rescue medication use, among children and adolescents with pediatric asthma.

DETAILED DESCRIPTION:
The primary study objective is to measure the effectiveness of using an innovative tracking system (CareTRx) for the self-management of asthma, including daily and rescue medication use, among children with asthma. The study objectives will be achieved using a pre-post design for the participants. The investigators aim to enroll at least 26 participants for a 3-month intervention period. With this pilot study, the investigators hope to examine the impact of self-management behaviors on health outcomes including asthma symptoms and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

1. Youth with a primary diagnosis of persistent asthma according by NHLBI criteria
2. Females or males between the ages of 6-17 years of age
3. Youth or caregiver must have an Android smart phone with operating system 4.3 or above and data plan for the duration of the study period

Exclusion Criteria:

1. Youth with other cardiac, pulmonary, or neuromuscular disorders that impact breathing
2. Youth with documented developmental delays or impairments that would interfere with ability to use CareTRx system

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, MD, MS, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] U.S. Department of Health and Human Services. Healthy People 2010: Understanding and Improving Health. 2nd ed. Washington DC: U.S. Government Printing Office; 2000.
- [Background] Forrest CB, Starfield B, Riley AW, Kang M. The impact of asthma on the health status of adolescents. Pediatrics. 1997 Feb;99(2):E1. doi: 10.1542/peds.99.2.e1. PMID 9099758
- [Background] Centers for Disease Control and Prevention (CDC). Self-reported asthma among high school students--United States, 2003. MMWR Morb Mortal Wkly Rep. 2005 Aug 12;54(31):765-7. PMID 16094284
- [Background] Akinbami LJ, Schoendorf KC. Trends in childhood asthma: prevalence, health care utilization, and mortality. Pediatrics. 2002 Aug;110(2 Pt 1):315-22. doi: 10.1542/peds.110.2.315. PMID 12165584
- [Background] National Asthma Education and Prevention Program. Expert Panel Report II: guidelines for the diagnosis and management of asthma. Bethesda, MD: National Institutes of Health; 1997
- [Background] Rapoff, MA. Adherence to pediatric medical regimens, 2nd ed. 2010; New York: Springer
- [Background] DiMatteo MR, Giordani PJ, Lepper HS, Croghan TW. Patient adherence and medical treatment outcomes: a meta-analysis. Med Care. 2002 Sep;40(9):794-811. doi: 10.1097/00005650-200209000-00009. PMID 12218770
- [Background] Halterman JS, Aligne CA, Auinger P, McBride JT, Szilagyi PG. Inadequate therapy for asthma among children in the United States. Pediatrics. 2000 Jan;105(1 Pt 3):272-6. PMID 10617735
- [Background] Blaschke TF, Osterberg L, Vrijens B, Urquhart J. Adherence to medications: insights arising from studies on the unreliable link between prescribed and actual drug dosing histories. Annu Rev Pharmacol Toxicol. 2012;52:275-301. doi: 10.1146/annurev-pharmtox-011711-113247. Epub 2011 Sep 19. PMID 21942628
- [Background] Palermo TM, Wilson AC. eHealth applications in pediatric psychology. In MC Roberts,RG Steele (Eds.), Handbook of pediatric psychology (4th ed., pp. 227-237). 2009. New York: Guilford
- [Background] Atienza AA, Stone AA, Shiffman S, Nebeling L. Introduction. In AA Stone, S Shiffman, AA Atienza, L Nebeling (Eds.), The science of real-time data capture: self-reports in health research. 2007; New York: Oxford
- [Background] Rapoff MA, Lootens CC, Tsai MS. Assessing adherence and barriers to adherence in pediatric asthma. Resp. Drug Deliv. 2012; 1-12
- [Background] Ingerski LM, Hente EA, Modi AC, Hommel KA. Electronic measurement of medication adherence in pediatric chronic illness: a review of measures. J Pediatr. 2011 Oct;159(4):528-34. doi: 10.1016/j.jpeds.2011.05.018. Epub 2011 Jul 1. No abstract available. PMID 21722917
- [Background] Dale O, Hagen KB. Despite technical problems personal digital assistants outperform pen and paper when collecting patient diary data. J Clin Epidemiol. 2007 Jan;60(1):8-17. doi: 10.1016/j.jclinepi.2006.04.005. Epub 2006 Aug 30. PMID 17161749
- [Background] Stone AA, Shiffman S, Schwartz JE, Broderick JE, Hufford MR. Patient compliance with paper and electronic diaries. Control Clin Trials. 2003 Apr;24(2):182-99. doi: 10.1016/s0197-2456(02)00320-3. PMID 12689739
- [Background] Palermo TM, Valenzuela D, Stork PP. A randomized trial of electronic versus paper pain diaries in children: impact on compliance, accuracy, and acceptability. Pain. 2004 Feb;107(3):213-219. doi: 10.1016/j.pain.2003.10.005. PMID 14736583
- [Background] Quittner AL, Modi AC, Lemanek KL, Ievers-Landis CE, Rapoff MA. Evidence-based assessment of adherence to medical treatments in pediatric psychology. J Pediatr Psychol. 2008 Oct;33(9):916-36; discussion 937-8. doi: 10.1093/jpepsy/jsm064. Epub 2007 Sep 10. PMID 17846042
- [Derived] Behrooz L, Dilley MA, Petty CR, Huffaker MF, Sheehan WJ, Phipatanakul W. The efficacy of a novel monitoring device on asthma control in children with asthma. Ann Allergy Asthma Immunol. 2020 Sep;125(3):352-354. doi: 10.1016/j.anai.2020.06.025. Epub 2020 Jun 20. No abstract available. PMID 32574599

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CareTRx Device
Started | 26
Completed | 24
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | CareTRx Device
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 9.1 [6 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 11
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Asthma control test [Mean (Standard Deviation); unit: units on a scale] — Asthma control test is a survey used to evaluate asthma control in patients. It includes 5 multiple questions that ask about how much of the time patient was having asthma symptoms. The higher the score the better asthma control. Lower scores especially less than 19 represent poor asthma control. each question has 5 answers. The total score is the sum of all the scores from 5 questions. the maximum score on the test is 25 which is excellent asthma control and the lowest is 0 which defines extremely poor asthma control.
  units on a scale | 20.6 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Daily Medication Compliance
Description: Total number participants who took their medication as planned will be measured. This will include measuring the number of participants with medication compliance who take their medications as planned based on the data from the monitoring device.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- CareTRx Device: All eligible participants will receive CareTRx device for control inhaler as well as the application downloaded to their Android phone. CareTRx is a novel monitoring device that can be applied to most MDI (meter dose inhaler) device and leverages mobile and cloud computing to objectively assess and provide information to patients and providers around medication adherence and disease control in pediatric asthma. The information will then be loaded to phone app.
  All data in the table represent values collected during the study and no placeholder values were used.
Arm/Group | CareTRx Device
Number analyzed (Participants) | 24
Participants | 24

2. Primary Outcome: Number of Participants With Rescue Inhaler Use
Description: Total number participants with rescue inhaler use throughout the course of the study.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- CareTRx Device: All eligible participants will receive CareTRx device for rescue inhaler as well as the application downloaded to their Android phone. CareTRx is a novel monitoring device that can be applied to most MDI (meter dose inhaler) device and leverages mobile and cloud computing to objectively assess and provide information to patients and providers around medication adherence and disease control in pediatric asthma. The information will then be loaded to phone app.
  All data in the table represent values collected during the study and no placeholder values were used.
Arm/Group | CareTRx Device
Number analyzed (Participants) | 24
Participants | 24

3. Secondary Outcome: Asthma Symptoms
Description: Asthma symptom control as a measure of effectiveness of self-management behavior on asthma control, measured by Asthma Control Test (ACT). Asthma control test is a survey used to evaluate asthma control in patients. It includes 5 multiple questions that ask about how much of the time patient was having asthma symptoms. The higher the score the better asthma control. Lower scores especially less than 19 represent poor asthma control. each question has 5 answers. The total score is the sum of all the scores from 5 questions. the maximum score on the test is 25 which is excellent asthma control and the lowest is 0 which defines extremely poor asthma control.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CareTRx Device
Number analyzed (Participants) | 24
units on a scale | 21.6 (3.9)

4. Secondary Outcome: Forced Expiratory Volume
Description: Forced expiratory volume measured in liters is the volume of air which can be forcibly exhaled from the lungs in the first second of a forced expiration and helps with evaluation of asthma control. FEV1 was only measure at baseline to assess the participants asthma status at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | CareTRx Device
Number analyzed (Participants) | 24
liters | 1.56 (0.62)

ADVERSE EVENTS:
Arm/Group | CareTRx Device
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No